CLINICAL TRIAL: NCT03001388
Title: Longitudinal Assessment of Transient Elastography in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ELASTIC-CF; U01DK062456 (NIH)
Record Dates: First submitted 2016-11-18; First posted 2016-12-23 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis Liver Disease
Keywords: Cystic Fibrosis Liver Disease; Pancreatic insufficiency; Cystic Fibrosis; Transient Elastography
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transient Elastography (TE) — Participants enrolled in Cystic Fibrosis Liver Disease Network (CFLD NET)Prediction by Ultrasound of the Risk of Hepatic Cirrhosis in Cystic Fibrosis (PUSH) study in longitudinal follow up at centers with Fibroscan available (currently 8/11 centers)

SUMMARY:
To determine if transient elastography (TE), when combined with ultrasound (US) pattern characterization can improve the prediction of progression to a nodular pattern on US.

To confirm the feasibility of obtaining TE measurements in children with Cystic Fibrosis (CF) To prospectively assess whether TE data are associated with conventional laboratory markers of hepatic fibrosis To determine the variability of TE measurements taken at different sites in the same patient

DETAILED DESCRIPTION:
A noninvasive assessment of hepatic fibrosis is desperately needed to advance the care of children with CF significant liver disease and to provide for measurements during clinical trials. That global assessment might serve as both a predictor/descriptor of disease course but also as a critical biomarker for clinical research. FibroScan® measurement of liver stiffness has great potential to fill this void. The underlying hypothesis of this proposal is that elastography in addition to US can improved the prediction of the development of a nodular liver on US and development of portal hypertension over time in children and young adults with CF.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in CFLD NET PUSH study in longitudinal follow up at centers with Fibroscan available (currently 8/11 centers)
* Entry criteria for that study were:
* CF as determined by sweat chloride >60 meq/l
* Pancreatic insufficiency
* Age 3-12 years old at entry
* For entry into the longitudinal follow up subjects were in one of two groups

  * A screening US pattern of nodular liver (CIR), heterogeneous increased echogenicity (HTG) or homogeneous increased echogenicity (HMG)
  * A screening US pattern of normal (NL) matched to a HTG subject (2 NL:1HTG) by age, center and pseudomonas status

Exclusion Criteria:

* Exited from the PUSH Study
* Unable / unwilling to sign consent

Ages: 6 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants enrolled in CFLD NET PUSH study in longitudinal follow up at centers with Fibroscan available (currently 8/11 centers) All racial and ethnic groups will be included.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Liver Stiffness Measurement (LSM) obtained via transient elastography using FibroScanTM | Baseline
  Liver stiffness" quantifies liver fibrosis and is measured in kPa (median of 10 subsequent valid measurements and are deemed acceptable if the ratio of interquartile range and median is <30% and success rate is >60%, meaning 10 valid measurements are obtained within 16 attempts).
Liver Stiffness Measurement (LSM) obtained via transient elastography using FibroScanTM | Year 1
  Liver stiffness" quantifies liver fibrosis and is measured in kPa (median of 10 subsequent valid measurements and are deemed acceptable if the ratio of interquartile range and median is <30% and success rate is >60%, meaning 10 valid measurements are obtained within 16 attempts).
Liver Stiffness Measurement (LSM) obtained via transient elastography using FibroScanTM | Year 2
  Liver stiffness" quantifies liver fibrosis and is measured in kPa (median of 10 subsequent

SECONDARY OUTCOMES:
Liver steatosis obtained via transient elastography | Baseline, Year 1, Year 2
  Controlled Attenuation Parameter (CAP)" quantifies liver steatosis and is measured in dB
Comparison of liver stiffness and liver steatosis measurements at each time point to grayscale ultrasound grades | Baseline, Year 1 and Year 2
  Grayscale ultrasound grades will be obtained from the parent study (PUSH: Clinical Trials: NCT01144507)
Comparison of liver stiffness and liver steatosis measurements at each time point to clinical findings of portal hypertension | Baseline, Year 1 and Year 2
  Grayscale ultrasound grades will be obtained from the parent study (PUSH: Clinical Trials: NCT01144507)

OTHER OUTCOMES:
Invalid measurements and success rate on liver stiffness and liver steatosis measurements | Baseline, Year 1 and Year 2
Inter quartile range (IQR) (kPa or dB/m) of all valid measurements within the examination | Baseline, Year 1 and Year 2
  To reflect the dispersion of stiffness and steatosis
IQR/median ratio of all valid measurements within the examination | Baseline, Year 1 and Year 2
  This quantity should remain as low as possible to ensure reliable results (goal < 30%)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (7):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye W, Leung DH, Molleston JP, Ling SC, Murray KF, Nicholas JL, Huang S, Karmazyn BW, Harned RK, Masand P, Alazraki AL, Navarro OM, Otto RK, Palermo JJ, Towbin AJ, Alonso EM, Karnsakul WW, Jane Schwarzenberg S, Seidel GF, Siegel M, Magee JC, Narkewicz MR, Jay Freeman A. Association Between Transient Elastography and Controlled Attenuated Parameter and Liver Ultrasound in Children With Cystic Fibrosis. Hepatol Commun. 2021 May 13;5(8):1362-1372. doi: 10.1002/hep4.1719. eCollection 2021 Aug. PMID 34430781
- See also: ChiLDReN Website — https://childrennetwork.org